CLINICAL TRIAL: NCT04262843
Title: Phase II Study of Evaluating the Efficacy of Total Marrow and Lymphoid Irradiation (TMLI) as the Conditioning Regimen for HLA-Haploidentical Hematopoietic Cell Transplantation in Patients With Myelodysplasia or Acute Leukemia
Brief Title: Total Marrow and Lymphoid Irradiation as Conditioning Regimen Before Hematopoietic Cell Transplantation in Patients With Myelodysplastic Syndrome or Acute Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19518; NCI-2019-08984 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19518 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2020-02-03; First posted 2020-02-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; High Risk Myelodysplastic Syndrome; Myelodysplastic Syndrome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Granulocyte Colony-Stimulating Factor; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Radiotherapy, Intensity-Modulated; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (fludarabine, TMLI, HCT, cyclophosphamide) (Experimental): CONDITIONING: Patients receive fludarabine IV QD on days -7 to -5, and undergo TMLI BID on days -4 to 0 in the absence of disease progression or unacceptable toxicity.
  TRANSPLANT: Patients undergo hematopoietic cell transplantation on day 0.
  GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV QD on days 3-4 in the absence of disease progression or unacceptable toxicity. Beginning on day 5, patients also receive granulocyte colony stimulating factor and tacrolimus/mycophenolate mofetil per institutional standard.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Fludarabine Phosphate; Biological: Granulocyte Colony-Stimulating Factor; Procedure: Hematopoietic Cell Transplantation; Procedure: Intensity-Modulated Radiation Therapy; Drug: Mycophenolate Mofetil; Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Biological: Granulocyte Colony-Stimulating Factor — Growth factor therapy
  Other Names: Colony Stimulating Factor 3; Colony-Stimulating Factor (Granulocyte); Colony-Stimulating Factor 3; CSF3; G CSF; G-CSF; Granulocyte Colony Stimulating Factor; Pluripoietin
Procedure: Hematopoietic Cell Transplantation — Undergo hematopoietic cell transplantation
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; Stem Cell Transplant; stem cell transplantation
Procedure: Intensity-Modulated Radiation Therapy — Undergo TMLI
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Drug: Mycophenolate Mofetil — Immunosuppressive therapy
  Other Names: Cellcept; MMF
Drug: Tacrolimus — Immunosuppressive therapy
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This phase II trial studies how well total marrow and lymphoid irradiation works as a conditioning regimen before hematopoietic cell transplantation in patients with myelodysplastic syndrome or acute leukemia. Total body irradiation can lower the relapse rate but has some fatal side effects such as irreversible damage to normal internal organs and graft-versus-host disease (a complication after transplantation in which donor's immune cells recognize the host as foreign and attack the recipient's tissues). Total body irradiation is a form of radiotherapy that involves irradiating the patient's entire body in an attempt to suppress the immune system, prevent rejection of the transplanted bone marrow and/or stem cells and to wipe out any remaining cancer cells. Intensity-modulated radiation therapy (IMRT) is a more recently developed method of delivering radiation. Total marrow and lymphoid irradiation is a method of using IMRT to direct radiation to the bone marrow. Total marrow and lymphoid irradiation may allow a greater dose of radiation to be delivered to the bone marrow as a preparative regimen before hematopoietic cell transplant while causing less side effects to normal organs than standard total body irradiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the efficacy of the haploidentical hematopoietic cell transplantation (haploHCT) total marrow and lymphoid organ irradiation (TMLI), with high dose post-transplant cyclophosphamide (PTCy) as graft-versus host disease (GvHD) prophylaxis, as assessed by 1-year graft versus (vs) host disease-free relapse-free survival (GRFS) rate in each arm (Arm A: patients with acute myeloid leukemia [AML] or myelodysplastic syndrome [MDS] and Arm B: Patients with acute lymphoblastic leukemia [ALL]).

SECONDARY OBJECTIVES:

I. Estimate overall survival (OS), cumulative incidences of relapse/disease progression, and non-relapse mortality (NRM) in each arm at 100 days, and 1 year post-transplant.

II. Estimate rate of relapse and non-relapse mortality (NRM) at 1 year post-transplant.

III. Estimate rates of acute and chronic GvHD, infections, complete remission and neutrophil recovery.

IV. Describe and characterize cytokine release syndrome (CRS) post-haploidentical HCT with TMLI as conditioning regimen and PTCy as GvHD prophylaxis as assessed by incidence, frequency and severity.

V. Further evaluate the safety of this regimen by assessing:

Va. Adverse events: type, frequency, severity, attribution, time course, duration.

Vb. Complications: including acute/chronic GVHD, infection and delayed engraftment.

EXPLORATORY OBJECTIVES:

I. Characterize minimal residual disease from bone marrow aspirates and investigate the possible association between TMLI-based regimen and patient's disease status.

II. Describe the kinetics of immune cell recovery. III. Describe the kinetics of serum pro-inflammatory cytokines and GvHD biomarkers.

IV. Longitudinal and spatial assessment of TMLI effect on bone marrow environment.

V. Cellular and molecular assessment of TMLI effect on bone marrow environment and TMLI effect on the engraftment and disease relapse.

OUTLINE:

CONDITIONING: Patients receive fludarabine intravenously (IV) once daily (QD) on days -7 to -5, and undergo TMLI twice daily (BID) on days -4 to 0 in the absence of disease progression or unacceptable toxicity.

TRANSPLANT: Patients undergo hematopoietic cell transplantation on day 0.

GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV QD on days 3-4 in the absence of disease progression or unacceptable toxicity. Beginning on day 5, patients also receive granulocyte colony stimulating factor and tacrolimus/mycophenolate mofetil per institutional standard.

After completion of study treatment, patients are followed up twice weekly for the first 100 days post-transplant, twice monthly until 6 months post-transplant, monthly until patient discontinues immunosuppressive therapy, and then yearly for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Karnofsky performance status >= 70
* Histologically confirmed diagnosis of one the following:

  * Patients with acute myelogenous leukemia

    * In first complete remission (CR1) with intermediate or poor risk cytogenetics according to National Comprehensive Cancer Network (NCCN) guidelines for acute myeloid leukemia (AML) or European LeukemiaNet (ELN) 2017
    * In second complete remission (CR2) or third complete remission (CR3)
    * Patients with chemosensitive active disease
  * Patients with acute lymphocytic leukemia

    * In CR1 with poor risk cytogenetics:
  * For adults according to NCCN guidelines for acute lymphoblastic leukemia (ALL): Patients older than 40 year of age; with high white blood cell count (WBC) at diagnosis (>= 30,000 for B lineage or >= 50,000 for T lineage), or with high risk cytogenetics including: hypoploidy (< 44 chromosomes); t(v;11q23): MLL rearranged; t(9;22) (q34;q11.2); complex cytogenetics (5 or more chromosomal abnormalities)
  * For pediatrics t(9;22), iAMP21loss of 13q, and abnormal 17p

    * In CR2 or CR3
    * Patients with chemosensitive active disease
  * Myelodysplastic syndrome in high-intermediate (int-2) and high risk categories by International Prognostic Scoring System (IPSS) or revised (R)-IPSS
* Total bilirubin =< 2 X upper limit of normal (ULN) (unless has Gilbert's disease) (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Creatinine clearance of >= 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Ejection fraction measured by echocardiogram or multigated acquisition scan (MUGA) >= 50% (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* If able to perform pulmonary function tests: forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and carbon monoxide diffusing capability test (DLCO) (diffusion capacity) >= 50% of predicted (corrected for hemoglobin). If unable to perform pulmonary function tests: oxygen (O2) saturation > 92% on room air

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR]) (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note: Infectious disease testing to be performed within 28 days prior to Day 1 of protocol therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* The recipient must have a related donor genotypically human leukocyte antigen (HLA)-A, B,C and DRB1 loci haploidentical to the recipient
* No HLA matched sibling or matched unrelated donor is available
* Patients should be off all previous intensive therapy, chemotherapy or radiotherapy for 3 weeks prior to commencing therapy on this study

  * (NOTE: Low dose chemotherapy or maintenance chemotherapy given within 7 days of planned study enrollment is permitted. These include: Hydroxyurea, 6-meraptopurine, oral methotrexate, vincristine, oral etoposide, and tyrosine kinase inhibitors [TKIs]. FLT-3 inhibitors such as sorafenib, crenolanib, midostaurin can also be given up to 3 days before conditioning regimen.)
* DONOR: The donor must be examined and have specific tests performed according to existing institutional guidelines to evaluate his/her candidacy as a donor including the following:
* DONOR: Age =< 60 years of age
* DONOR: For younger donors, no more than 20 mL bone marrow may be harvested per kg of donor body weight
* DONOR: Medical history and physical examination confirm good health status as defined by institutional standards
* DONOR: Seronegative for HIV Ag, HIV 1+2 Ab, HTLV I/II Ab, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) (IgM and IgG), HCV Ab, RPR for syphilis within 30 days of apheresis collection
* DONOR: Genotypically haploidentical as determined by HLA typing, preferably a nonmaternal HLA haploidentical relative due to data of high incidence of graft failure with use of maternal HLA haploidentical cells. Eligible donors include biological parents, siblings or half siblings, or children
* DONOR: Female donors of child-bearing potential must have a negative serum or urine beta-human chorionic gonadotropin (HCG) test within seven days of mobilization
* DONOR: The donor must have been informed of the investigational nature of this study and have signed a consent form in accordance with Federal Guidelines and the guidelines of the participating institution
* DONOR: Selection of a haploidentical donor will require absence of pre-existing donor-directed anti-HLA antibodies in the recipient

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active bacterial, viral or fungal infection
* Patient may not be receiving any other investigational agents or concurrent biological, intensive chemotherapy or radiation therapy for the previous three weeks from conditioning

  * (NOTE: Low dose chemotherapy or maintenance chemotherapy given within 7 days of planned study enrollment is permitted. These include: Hydroxyurea, 6-meraptopurine, oral methotrexate, vincristine, oral etoposide, and tyrosine kinase inhibitors [TKIs]. FLT-3 inhibitors such as sorafenib, crenolanib, midostaurin can also be given up to 3 days before conditioning regimen.)
* Herbal medications dependency
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* No intercurrent illness or other malignancy (other than non-melanoma skin cancer)
* Active infection requiring antibiotics
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Patients who had a prior autologous or allogeneic transplant
* Patients who had prior radiation therapy of more than 20% of bone marrow containing areas or to any area exceeding 2000 cGy
* Patients with HLA-matched or partially matched (7/8 or 8/8) related or fully matched unrelated donor available to donate
* Patients who have received more than 3 prior regimens, where the regimen intent was to induce remission
* Patients with treatment history including anti-CD33 monoclonal antibody therapy (e.g., SGN-CD33 or Mylotarg)
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)
* DONOR: Evidence of active infection
* DONOR: Medical or physical reason which makes the donor unlikely to tolerate or cooperate with growth factor therapy and leukapheresis
* DONOR: Factors which place the donor at increased risk for complications from leukapheresis or granulocyte colony-stimulating factor (G-CSF) therapy
* DONOR: HIV positive

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-06-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to day 100
  Evaluated using the Bearman scale and National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Graft-versus-host disease (GvHD) free relapse-free survival | Time from start of protocol therapy to grade 3-4 acute GvHD, chronic GvHD requiring systemic treatment, death, relapse/progression, or last follow-up, whichever comes first, assessed up to 2 years post-transplant

SECONDARY OUTCOMES:
Overall survival | Time from start of protocol therapy to death from any cause, or last follow-up, whichever comes first, assessed up to 2 years post-transplant
Relapse-free survival | Time from the start of protocol therapy to the date of death, disease relapse, or last follow-up, whichever comes first, assessed up to 2 years post-transplant.]
Time to relapse/progression | Time from the start of protocol therapy to death, disease relapse or progression, or last follow-up, whichever comes first, assessed up to 2 years post-transplant
Non-relapse mortality | Time from start of therapy until non-disease related death, or last follow-up, whichever comes first, assessed up to 2 years post-transplant
Incidence of adverse events that meet grade 3, 4, or 5 per CTCAE version 5.0 | From day -9 to day -1, from day 0 to day 30, and day 31 to day 100 post-transplant
Incidence of acute GvHD of grades 2-4 and 3-4 | From date of stem cell infusion to documented/biopsy proven acute GVHD onset date (within the first 100 days post-transplant)
Incidence of chronic GvHD | From approximately 80-100 days post-transplant to the documented/biopsy proven chronic GvHD onset date
Incidence of infection | From day 0 to day 100 post-transplant
Complete remission proportion | At day 30
Rate of neutrophil recovery | Up to 2 years
  Measured from stem cell infusion to the first to three consecutive days with neutrophil count greater than 0.5 x 10^9/l.
Incidence of cytokine release syndrome | Up to 2 years
  Defined and graded per American Society for Transplantation and Cellular Therapy (ASTCT) criteria.

OTHER OUTCOMES:
Minimal residual disease | At day 30, 100, and 180 days, and 1 year post-transplant
  Assessed from bone marrow aspirates.
Immune cell recovery | Up to 2 years
  Immunophenotyping with lymphocyte subsets by flow cytometry, including but not limited to the following cell markers: CD4, CD8, CD56, CD16, etc.
GvHD biomarker analysis | Up to 2 years
  Will be done by standard enzyme-linked immunosorbent (ELISA) assays.
Pro-inflammatory cytokine analysis | Up to 2 years
  Will be done using standard ELISA assays.
Effect of TMLI on bone marrow environment | Up to 2 years
  Longitudinal assessment swill be done by dual energy computed tomography (DECT), water-fat magnetic resonance imaging (wfMRI) imaging. Biological assessment of bone marrow samples will be done by flow cytometry, colony forming assay, and immunohistochemistry studies.

CONTACTS AND LOCATIONS:
Overall Officials: Monzr M Al Malki, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States